CLINICAL TRIAL: NCT01628094
Title: Randomized, Open-Label, Multicenter Study of Safety, Efficacy, and Tolerability of the Combination of RO5466731, RO5190591, Ritonavir, and Copegus With or Without RO5024048 in HCV Genotype 1 Infected Patients Who Are Either Treatment Naïve or Null Responders to Previous Interferon-Based Treatment
Brief Title: ANNAPURNA: A Study of The Combination of RO5466731, RO5190591, Ritonavir and Copegus (Ribavirin) With or Without RO5024048 in Patients With Chronic Hepatitis C Who Are Either Treatment-Naïve or Have Previously Experienced a Null Response to Interferon-Based Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP28266; 2012-000638-21 (EudraCT Number)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; Ritonavir

ARMS (6):
- A: GT1a 3DAA (Experimental): including RO5466731, RO5190591, ritonavir, ribavirin [Copegus] and RO5024048
  Interventions: Drug: RO5024048; Drug: RO5190591; Drug: RO5466731; Drug: ribavirin [Copegus]; Drug: ritonavir
- B: GT1a 3DAA (Experimental): including RO5466731, RO5190591, ritonavir, ribavirin [Copegus] and RO5024048
  Interventions: Drug: RO5024048; Drug: RO5190591; Drug: RO5466731; Drug: ribavirin [Copegus]; Drug: ritonavir
- C: GT1a 2DAA (Experimental): including RO5466731, RO5190591, ritonavir and ribavirin [Copegus]
  Interventions: Drug: RO5190591; Drug: RO5466731; Drug: ribavirin [Copegus]; Drug: ritonavir
- D: GT1b 3DAA (Experimental): including RO5466731, RO5190591, ritonavir, ribavirin [Copegus] and RO5024048
  Interventions: Drug: RO5024048; Drug: RO5190591; Drug: RO5466731; Drug: ribavirin [Copegus]; Drug: ritonavir
- E: GT1b 2DAA (Experimental): including RO54664731, RO5190591, ritonavir and ribavirin [Copegus]
  Interventions: Drug: RO5190591; Drug: RO5466731; Drug: ribavirin [Copegus]; Drug: ritonavir
- Part II (Experimental)
  Interventions: Drug: RO5024048; Drug: RO5190591; Drug: RO5466731; Drug: ribavirin [Copegus]; Drug: ritonavir

INTERVENTIONS:
Drug: RO5024048
  Arms: A: GT1a 3DAA; B: GT1a 3DAA; D: GT1b 3DAA; Part II
Drug: RO5190591
Drug: RO5466731
Drug: ribavirin [Copegus]
Drug: ritonavir

SUMMARY:
This randomized, open-label, multicenter study will evaluate the safety , efficacy and tolerability of the combination treatment RO5466731, RO5190591, ritonavir and Copegus (ribavirin) with or without RO5024048 in patients with chronic hepatitis C genotype 1. In Part 1, treatment-naïve patients will be randomized to receive treatment with RO5466731, RO5190591 plus ritonavir, and Copegus, with or without RO5024048. In Part 2, further treatment-naïve patients will receive a successful regimen from Part 1, or a reduced intensity regimen, and patients who have previously experienced null response to interferon-based treatment will be added to the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis C genotype 1 of >/= 6 months duration at screening
* Part 1 and Part 2: Naïve to treatment with interferon (pegylated or non-pegylated). Patients who have participated in studies investigating a direct-acting antiviral agent with or without interferon are excluded
* Part 2: Treatment experienced patients having a previous null response to treatment with interferon containing regimen
* Liver biopsy or non-invasive (e.g. Fibroscan) evaluation in the past 24 calendar months showing absence of cirrhosis or incomplete/transition to cirrhosis
* Body mass index (BMI) 18 to 35 kg/m2 inclusive and body weight >/= 45 kg

Exclusion Criteria:

* Pregnant or lactating women or males with female partners who are pregnant or lactating
* Decompensated liver disease or impaired liver function (as defined by protocol)
* Cirrhosis or incomplete/transition to cirrhosis
* Non- hepatitis C chronic liver disease
* Positive for hepatitis B or HIV infection
* History of pre-existing renal disease
* History of severe cardiac disease
* History of neoplastic disease within the last 5 years, except for localized or in situ carcinoma of the skin
* History of drug abuse within the last year; history of cannabinoid use is not excluded
* Evidence of alcohol abuse within 1 year of screening and consumption of more than 2 units of alcohol per day
* Medical condition that requires use of systemic corticosteroids
* Received warfarin or other anticoagulants during the 21 days immediately prior to screening or is expected to require warfarin or other anticoagulants during the study
* Anticipated use or need for significant medical treatment during the study or use of concomitant medications or nutrients that are excluded by protocol (e.g. drugs that are contraindicated with ritonavir, hormonal methods of contraception)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (defined as undetectable serum HCV RNA) 12 weeks after end of treatment | approximately 20 months
Safety: Incidence of adverse events | approximately 20 months

SECONDARY OUTCOMES:
Antiviral activity: Change in serum HCV RNA levels | from baseline to 24 weeks after end of treatment
Pharmacokinetics in coadministration: Area under the concentration-time curve (AUC) | Pre-dose Weeks 1, 2, 3, 4, 6, 10, and 12 and up to 12 hours post-dose Weeks 1, and 4 or 3 and 6
HCV drug resistance | approximately 20 months
Quality of life: Short-Form 36v2/Brief Fatigue Inventory questionnaires | approximately 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (14):
  - La Jolla, California
  - Englewood, Colorado
  - South Miami, Florida
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Kansas City, Kansas
  - Detroit, Michigan
  - Saint Louise, Missouri
  - Asheville, North Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Vancouver, Washington
- Australia (5):
  - Kingswood, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - Herston, Queensland
  - Parkville, Victoria
- Germany (4):
  - Berlin
  - Frankfurt am Main
  - Hamburg
  - Hanover
- New Zealand (3):
  - Dunedin
  - Grafton
  - Hamilton
- Poland (4):
  - Bialystok
  - Chorzów
  - Lodz
  - Mysłowice

REFERENCES:
- [Derived] Jensen DM, Brunda M, Elston R, Gane EJ, George J, Glavini K, Hammond JM, Le Pogam S, Najera I, Passe S, Piekarska A, Rodriguez I, Zeuzem S, Chu T; ANNAPURNA study investigators. Interferon-free regimens containing setrobuvir for patients with genotype 1 chronic hepatitis C: a randomized, multicenter study. Liver Int. 2016 Apr;36(4):505-14. doi: 10.1111/liv.12997. Epub 2015 Dec 12. PMID 26519669